CLINICAL TRIAL: NCT03096613
Title: Efficacy and Safety of Levothyroxine (L-T4) Replacement on Exercise Capability in Chronic Systolic Heart Failure Patients With Subclinical Hypothyroidism: A 24-week, Multi-center, Open Label, Randomized, Parallel Group Trial
Brief Title: Thyroid Hormone Replacement for Subclinical Hypothyroidism and Chronic Heart Failure (ThyroHeart-CHF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: The Luhe Teaching Hospital of the Capital Medical University (Other); Tianjin Medical University Second Hospital (Other); The First Hospital of Hebei Medical University (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Professor, chief physician, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-798
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Subclinical Hypothyroidism
Keywords: heart failure; Subclinical Hypothyroidism; levothyroxine; 6-minute walk test
MeSH Terms: conditions — Heart Failure | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levothyroxine group (Experimental): The patients allocated to levothyroxine group receive levothyroxine with a starting dose of 12.5ug.
  Interventions: Drug: Levothyroxine
- Standard therapy group (No Intervention): The patients in this group receive standard therapy in consistent with the local clinical practice.

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine is used to normalize the thyroid hormone level of patients allocated to levothyroxine.
  Other Names: Euthyrox
  Arms: Levothyroxine group

SUMMARY:
Based on accumulating evidence showing that hypothyroid status is associated with poor prognosis among heart failure (HF) patients, the study is designed to evaluate whether replacement treatment with levothyroxine could have beneficial effects on patients with HF and subclinical hypothyroidism. The study is a prospective, randomized, parallel-group trial to assess the efficacy and safety of levothyroxine replacement on evidence-based HF standard therapy in stable chronic heart failure patients with subclinical hypothyroidism.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine whether the 24-week L-T4 replacement therapy, as an adjunct to standard treatment, would improve exercise capability in chronic systolic heart failure patients with subclinical hypothyroidism compared to the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, male or female.
* Systolic heart failure with New York Heart Association (NYHA) class II-III.
* Left ventricular ejection fraction (LVEF) less than 40% by echocardiography during screening and randomization.
* SCH (TSH: upper limits of normal (ULN) -10mIU/L, and FT4 level within reference range).
* Having received standard HF therapy for at least 2 weeks, having reached target dose or max tolerable dose.
* Provided informed consent.

Exclusion Criteria:

* Acute heart failure or acute exacerbation of chronic heart failure within the past 2 weeks.
* Scheduled cardiac resynchronization therapy or heart transplantation.
* History of malignant tumor or life expectancy under 12 months.
* Already on medications that may affect thyroid function (L-T4, carbimazole, propylthiouracil, amiodarone, lithium).
* Pregnancy and lactation period.
* Participation in another clinical trial within the past 30 days.
* Contraindication or intolerance to evidence-based therapy for CHF, such as beta-blocker, angiotensin-converting enzyme inhibitor or angiotensin receptor blocker.
* Known hypersensitivity to the trial treatment(s) or diluents (when applicable), including placebo or other comparator drug(s).
* Untreated adrenal insufficiency.
* Untreated pituitary insufficiency.
* Untreated thyrotoxicosis.
* Treatment with levothyroxine must not be initiated in patients with acute myocardial infarction, acute myocarditis, or acute pancarditis.
* Severe renal dysfunction (eGFR≤30 ml/min/1.73m2).
* Significant hepatic impairment (Serum GPT > 120 U/L).
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Distance difference of Six-minute Walk Test (6MWT) between week 24 and baseline | Within 6 months of patient enrolled

SECONDARY OUTCOMES:
Difference of the plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP) level between week 24 and baseline | Within 6 months of patient enrolled
Change in NYHA classification between week 24 and baseline. | Within 6 months of patient enrolled
Composite of cardiovascular death or heart failure re-hospitalization during the 24 weeks treatment | Within 6 months of patient enrolled
Composite of cardiovascular death, re-hospitalization for cardiovascular disease, severe arrhythmia, and stroke during the 24 weeks treatment | Within 6 months of patient enrolled
Difference of echocardiographic and cardiac magnetic resonance imaging measures between week 24 and baseline | Within 6 months of patient enrolled
Difference of MLHFQ between week 24 and baseline | Within 6 months of patient enrolled
Difference of serum lipid profiles between week 24 and baseline | Within 6 months of patient enrolled
Adverse events | Within 6 months of patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang W, Zhang X, Gao J, Meng X, Wang J, Zhang K, Chen J, Qi J, Shao C, Tang YD. Effects of levothyroxine in subclinical hypothyroidism and heart failure with reduced ejection fraction: An open-label randomized trial. Cell Rep Med. 2024 Apr 16;5(4):101473. doi: 10.1016/j.xcrm.2024.101473. Epub 2024 Mar 26. PMID 38537636
- [Derived] Zhang X, Wang WY, Zhang K, Tian J, Zheng JL, Chen J, An SM, Wang SY, Liu YP, Zhao Y, Wang JJ, Yang M, Tang YD. Efficacy and safety of levothyroxine (L-T4) replacement on the exercise capability in chronic systolic heart failure patients with subclinical hypothyroidism: Study protocol for a multi-center, open label, randomized, parallel group trial (ThyroHeart-CHF). Trials. 2019 Feb 19;20(1):143. doi: 10.1186/s13063-019-3219-5. PMID 30782213